CLINICAL TRIAL: NCT06428058
Title: Evaluating the Effects of Reproductive Health Training on Provider Behavior
Acronym: THP-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01HD092655 (NIH)
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Health Knowledge, Attitudes, Practice; Training
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Testing of an Afrocentric sexual health curriculum for Midwifery, Nursing and Medical Students.
Who Masked: Outcomes Assessor
Masking Description: A randomized, controlled, single blinded trial, stratified by health profession, of the intervention vs waitlist control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive Sexual Health Curriculum (Experimental): Participants received a four-day comprehensive sexual health curriculum tailored for Africa.
  Interventions: Behavioral: Comprehensive sexual health curriculum
- Waitlist Control (No Intervention): Participants in this arm completed a follow-up survey and scheduled to receive the intervention after the end of the trial.

INTERVENTIONS:
Behavioral: Comprehensive sexual health curriculum — This is a randomized, controlled, single blinded, trial, stratified by health profession, of the intervention versus waitlist control assessing the effects on sexual health knowledge, attitudes, and sexual history and counseling skills at medium (6-) and long-term (12 and 24 months) follow-up. At the end of the intervention as compared with waitlist controls.
  The intervention was a 4-day, Afrocentric, comprehensive sexual health curriculum. Tanzanian faculty wrote the curriculum in English and Kiswahili to address the most common sexual health challenges clinicians experience in Tanzania. The 4-day curriculum covers sexual health across the lifespan, lesbian, gay, bisexual, and transgender (LGBT) and sexual violence, clinical skills training, ethics, and community resources and cultural considerations.
  Arms: Comprehensive Sexual Health Curriculum

SUMMARY:
The goal of this randomized, controlled, single blinded trial is to evaluate the medium to long-term effects of an Afrocentric sexual health curriculum on health professional students' knowledge, attitudes, and clinical skills in providing sexual health in Tanzania.

DETAILED DESCRIPTION:
All enrollees will be health students at MUHAS recruited through announcements in class, flyers on student noticeboards, and email. Students who are interested in learning more about the study can do so by asking questions of the recruiting faculty member, by going to, telephoning, or emailing the study office (at MUHAS). Students can also visit the study website. In addition, all students who contact the office will be given a copy of a flyer advertising the study and a copy of the consent documents to preview prior to participation. Students contacting the office by email will be sent electronic versions of the same documents.

Participants in Aim 1 are informed to schedule an appointment (in the month prior to the seminar) to complete a pre-evaluation. At the study site, participants complete pen and paper surveys, and are videotaped interviewing two standardized patients. Next, participants are randomized to either the intervention or waitlist control condition. Participants in the intervention will attend the 4-day sexual health seminar and complete a short post-test. In addition, at 6- and 12-month follow-up after the pre-test, participants in both arms complete surveys and two videotaped interviews (at each follow-up) and a final survey at 24-month follow-up. At the end of the study, participants assigned to the control condition can attend the seminar.

ELIGIBILITY:
Inclusion Criteria:

* A health student studying at MUHAS and verified by being registered as a pre-final year midwifery, nursing or medical student (or its equivalent).
* "Pre-final" year is defined as a student who is just about to enter year 3 of nursing, or year 4 of midwifery or medicine.
* Living or studying in Tanzania
* Experienced, operationalized as having worked at least 100 hours as a health worker in a clinic, hospital or community setting so students can discuss what happens in the clinical setting
* Able to speak English and Kiswahili.

Exclusion Criteria:

* Students who will not be able to attend all days of the seminar at their health institution or be on their campus for the follow-up.
* Students who express any reservations about attending (e.g., due to religious objections)
* Students who express a fear of violence due to attending (e.g., from a spouse or relative).
* Students who attended the sexual health seminar (e.g., during THP-1 or at another site). This is to prevent a student participating more than once.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2025-08-02 (Actual); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Sexual Health Knowledge Score | Baseline, 6-month follow-up, 12-month follow-up, and 24-month follow-up.
  Sexual health knowledge was assessed using 16 multichoice items created by the research team. The items covered female sexual health concerns (2 items), sexual development and masturbation (3 items), sexual orientation (3 items), sexual violence (3 items), sexuality in middle age (3 items), sexual history taking and sexual counseling (2 items). Total scores were used for analysis (maximum total score of 16). Participants get one point for every item answer correctly. Because there are 16 items in this section, participants can have a minimum total score of 0 and a maximum total score of 16. A higher score signifies better sexual health knowledge.
Change in Sexual Health Attitudes: Confidence in Ability to Discuss | Baseline, 6-month follow-up, 12-month follow-up, and 24-month follow-up.
  Confidence in their ability to discuss the sexual health of patients, and confidence in their ability to discuss their patients' sexual health concerns were assessed using the Sexual Health Education for Professionals Scale (SHEPS). This section consists of 37 items where participants rate their confidence from (1) very unconfident to (5) confident. Because there are 37 items in this section, participants can have a minimum total score of 37 and a maximum total score of 185. A higher value signifies better confidence in the ability to discuss sexual health topics.
Change in Sexual Health Attitudes: Confidence in Having Knowledge | Baseline, 6-month follow-up, 12-month follow-up, and 24-month follow-up.
  Confidence in their knowledge to assess the sexual health of patients, and confidence in their ability to discuss their patient's sexual health concerns were assessed using the Sexual Health Education for Professionals Scale (SHEPS). This section consists of 37 items where participants rate their confidence from (1) very unconfident to (5) confident. Because there are 37 items in this section, participants can have a minimum total score of 37 and a maximum total score of 185. A higher value signifies better confidence in having knowledge of sexual health topics.
Change in Sexual Counseling Skills: Interpersonal Communications | Baseline, 6-month follow-up, 12-month follow-up, and 24-month follow-up.
  Skills were assessed by faculty raters assessing two videos (per each time point) of student counseling blind to whether the participant was in the intervention or control group and whether the assessment was at baseline or follow-up. Each participant was rated on 10 items assessing their interpersonal communication (IC) abilities. Each item was on a 3-point scale (0=not done; 1=partially done; 2=done). The scale has a minimum score of 0 and a maximum score of 20 per video. The investigators aggregated scores for each time point by summing the two videos at each time point. Therefore, the minimum total score is 0 and the maximum total score is 40. A higher score value signifies better interpersonal communication skills.
Change in Sexual Counseling Skills: Medical History Taking | Baseline, 6-month follow-up, 12-month follow-up, and 24-month follow-up.
  Skills were assessed by faculty raters assessing the two videos (per time point) of student counseling blind to whether the participant was in the intervention or control group and whether the assessment was at baseline or follow-up. Medical history taking (MHT) was rated by six key pieces of information on a 2-point scale, where 0=not obtained information and 1=obtained information. The scale has a minimum score of 0 and a maximum score or 6 per video. The investigators aggregated scores for each time point by summing the two videos at each time point. Therefore, the minimum total score is 0 and the maximum total score is 12.
Change in Sexual Health Beliefs | Baseline, 6-month follow-up, 12-month follow-up, and 24-month follow-up.
  The SHEPS Attitudes section comprises 27 items. Participants rate their level of agreement (1=strongly agree; 5=strongly disagree), with 13 items being reverse coded. Because there are 27 items in this section, participants can have a minimum total score of 27 and a maximum total score of 135. Low scores correspond to "liberal" views and high scores correspond to "conservative" views.

CONTACTS AND LOCATIONS:
Overall Officials: B.R. Simon Rosser, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No
Only group data will be analyzed.